CLINICAL TRIAL: NCT01061671
Title: Prospective Randomized Placebo-Controlled Trial of SimvaSTATin in the Prevention of COPD Exacerbations (STATCOPE)
Brief Title: Simvastatin Therapy for Moderate and Severe COPD
Acronym: STATCOPE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 689; U10HL074424 (NIH)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Exacerbation; Lung function; Cardiovascular; Smoking; Statins; Simvastatin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking | interventions — Simvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- simvastatin (Active Comparator): 40 mgms of simvastatin daily
  Interventions: Drug: simvastatin
- placebo (Placebo Comparator): Matched placebo pill daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: simvastatin — 40 mgms of simvastatin daily
  Other Names: Zocor
  Arms: simvastatin
Drug: Placebo — Matched placebo pill daily
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
To determine the effect of daily administration of 40 mgms simvastatin taken for at least 12 months (range 12-36 months) on the frequency of exacerbations of chronic obstructive lung disease (COPD) in patients with moderate to severe COPD who are prone to exacerbations and do not have other indications for statin treatment.

DETAILED DESCRIPTION:
COPD exacerbation is a common complication that significantly contributes to the high morbidity, mortality and costs associated with COPD. COPD exacerbations are associated with heightened lung inflammation that may have systemic implications (e.g., peripheral muscle weakness, cognitive impairment, depression, stroke, acute coronary syndrome, and atherosclerosis). Statins are potent agents that significantly reduce vascular events in patients with increased risks due to prior cardiac or cerebral vascular events and elevated lipid profiles. Statins have pleiotropic effects that extend well beyond their lipid lowering effects and may be potent anti-inflammatory agents. Retrospective data conducted in COPD patients indicate that statin use is associated with markedly decreased rates of COPD hospitalization and stabilization of lung function. Decreases in mortality in COPD due to complications of flu-like illnesses and deaths due to cardiovascular events have also been reported. Inflammatory biomarkers (C-reactive protein and interleukin- 6) are reported to be elevated in moderate to severe COPD patients who are prone to exacerbations. Inflammatory biomarkers (C-reactive protein and interleukin- 6) are reported to be reduced by statin therapy in patients with hyperlipidemia and cardiovascular diseases. Treatments that can effectively lessen the prevalence and severity of COPD exacerbations are desperately needed

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 40-80 years of age.
2. Clinical diagnosis of at least moderate COPD as defined by the GOLD criteria:

   1. Postbronchodilator FEV1(forced expiratory volume at one second)/FVC(forced vital capacity) < 70%,
   2. Postbronchodilator FEV1 (forced expiratory volume at one second) < 80% predicted, with or without chronic symptoms (i.e., cough, sputum production).
3. Cigarette consumption of 10 pack-years or more. Patients may or may not be active smokers.
4. Must meet one or more of the following 4 conditions

   1. Be using supplemental oxygenate
   2. Receiving a course of systemic corticosteroids and/or antibiotics for respiratory problems in the past year,
   3. Visiting an Emergency Department for a COPD exacerbation within the past year, or
   4. Being hospitalized for a COPD (Chronic Obstructive Pulmonary Disease) exacerbation within the past year
5. Willingness to make return visits and availability by telephone for duration of study.
6. Free of active coronary disease
7. Subject with expected life expectancy > 36 months

Exclusion Criteria:

1. Patients who:

   1. are on statin drugs.
   2. should be on statins based on established risk stratification using the ATP-III (Adult Treatment Panel) to determine 10 year risk.
2. Documented history of active coronary heart disease, such as unstable angina, prior myocardial infarction, stroke, symptomatic peripheral vascular or carotid artery disease, or congestive heart failure within the past 3 months.
3. A diagnosis of asthma.
4. The presence of a diagnosis other than COPD that results in the patient being either medically unstable, or having a predicted life expectancy < 3 years.
5. Special patient groups: prisoners, pregnant women, institutionalized patients
6. Women who are at risk of becoming pregnant during the study (pre-menopausal) and who refuse to use acceptable birth control (hormone-based oral or barrier contraceptive) for the duration of the study.
7. Woman using estradiol compounds for contraception. Postmenopausal women on estradiol compounds for hormone replacement therapy will be allowed into the trial.
8. Participants otherwise meeting the inclusion criteria will not be enrolled until they are a minimum of four weeks from their most recent acute exacerbation.
9. A clinical diagnosis of bronchiectasis defined as production of > one-half cup of purulent sputum/day.
10. Participants using niacin, azole antifungals (itraconazole, ketoconazole, posaconazole), fibric acid derivatives, erythromycin, clarithromycin, telithromycin, diltiazem, amlodipine , ranolazine,HIV protease inhibitors (such as indinavir), amiodarone, gemfibrozil, cyclosporine, verapamil, danazol, nefazodone, and red yeast rice extracts are excluded
11. Active liver disease. Active liver disease is defined as ALT (alanine aminotransferase), AST (aspartate aminotransferase) as greater than 1.5 times the upper limit of normal.
12. Patients with renal failure defined by serum creatinine greater than 3mg/dl.
13. Alcoholism. Alcoholism is defined as > 35 drinks per week. A drink is defined as one bottle of beer, one 8-ounce glass of wine, or one ounce of hard liquor.
14. Hypersensitivity to HMG CoA (3-hydroxy-3-methylglutaryl-coenzyme A) reductase inhibitors. Hypersensitivity is defined as an allergic reaction to statin, prior history of myopathy, rhabdomyolysis or previous intolerance to statin use.
15. Participants drinking greater than 4 cups (1qt) of grapefruit juice per day.
16. Participants drinking greater than 3 cups of green tea per day.
17. Diabetics will be excluded. Diabetics are defined by:

1. A CURRENT physician diagnosis of diabetes OR 2. CURRENT use of diabetic meds OR 3. Elevated HbA1c > 6.5% 18. The discretion of the Principal Investigator that the potential participant will not be a reliable study subject to complete the study requirements.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Connett, PhD, Principal Investigator — University of Minnesota (Data Coordinating Center); Steven M Scharf, MD, PhD, Principal Investigator — University of Maryland, Baltimore; Mark Dransfield, MD, Principal Investigator — University of Alabama at Birmingham; George Washko, MD, Principal Investigator — Brigham and Women's Hospital Boston; Richard K Albert, MD, Principal Investigator — Denver Health Medical Center; Richard Casaburi, MD, PhD, Principal Investigator — Harbor-UCLA Research & Education Institute; Dennis E Niewoehner, MD, Principal Investigator — Minnesota Veterans Affairs Medical Center; Gerard J Criner, MD, Principal Investigator — Temple University Philadelphia; Frank Sciurba, MD, Principal Investigator — University of Pittsburgh; Stephen C Lazarus, MD, Principal Investigator — University of California at San Francisco; Fernando J Martinez, MD, Principal Investigator — University of Michigan; Don Sin, M.D., Principal Investigator — St. Paul's Hospital; Shawn Aaron, M.D., Principal Investigator — The Ottawa Hospital
Locations (51):
- United States (35):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Veteran's Administration Medical Center, Birmingham, Alabama
  - LA BioMed at Harbor-UCLA Medical Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois Health System, Chicago, Illinois
  - LSU Health, New Orleans, Louisiana
  - University of Maryland Baltimore, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Veteran's Administration Medical Center, Boston, Massachusetts
  - Reliant Medical Group, Worcester, Massachusetts
  - Veteran's Administration Medical Center, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Veteran's Administration Medical Center, Minneapolis, Minnesota
  - HealthPartners Research Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Lovelace Respiratory Research Institute, Albuquerque, New Mexico
  - Western New York Veterans Administration Healthcare System, Buffalo, New York
  - Duke University, Durham, North Carolina
  - Cincinnati VAMC, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Institute for Respiratory and Sleep, Langhorne, Pennsylvania
  - Temple University Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Pittsburgh VA Medical Center, Pittsburgh, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
- Canada (16):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Lion's Gate Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (Laval Hospital), Québec

REFERENCES:
- [Derived] Camac ER, Voelker H, Criner GJ; COPD Clinical Research Network and the Canadian Institutes of Health Research. Impact of COPD exacerbations leading to hospitalization on general and disease-specific quality of life. Respir Med. 2021 Sep;186:106526. doi: 10.1016/j.rmed.2021.106526. Epub 2021 Jun 29. PMID 34229290
- [Derived] Rao AK, Del Carpio-Cano F, Janapati S, Zhao H, Voelker H, Lu X, Criner G; NIH COPD Clinical Research Network, the Canadian Institute of Health Research Investigators. Effects of simvastatin on tissue factor pathway of blood coagulation in STATCOPE (Simvastatin in the prevention of COPD exacerbations) trial. J Thromb Haemost. 2021 Jul;19(7):1709-1717. doi: 10.1111/jth.15282. Epub 2021 Apr 12. PMID 33638931
- [Derived] Leitao Filho FS, Ra SW, Mattman A, Schellenberg RS, Criner GJ, Woodruff PG, Lazarus SC, Albert R, Connett JE, Han MK, Martinez FJ, Leung JM, Paul Man SF, Aaron SD, Reed RM, Sin DD; Canadian Respiratory Research Network (CRRN). Serum IgG subclass levels and risk of exacerbations and hospitalizations in patients with COPD. Respir Res. 2018 Feb 14;19(1):30. doi: 10.1186/s12931-018-0733-z. PMID 29444682
- [Derived] Brown KE, Sin DD, Voelker H, Connett JE, Niewoehner DE, Kunisaki KM; COPD Clinical Research Network. Serum bilirubin and the risk of chronic obstructive pulmonary disease exacerbations. Respir Res. 2017 Oct 24;18(1):179. doi: 10.1186/s12931-017-0664-0. PMID 29065885
- [Derived] Criner GJ, Connett JE, Aaron SD, Albert RK, Bailey WC, Casaburi R, Cooper JA Jr, Curtis JL, Dransfield MT, Han MK, Make B, Marchetti N, Martinez FJ, Niewoehner DE, Scanlon PD, Sciurba FC, Scharf SM, Sin DD, Voelker H, Washko GR, Woodruff PG, Lazarus SC; COPD Clinical Research Network; Canadian Institutes of Health Research. Simvastatin for the prevention of exacerbations in moderate-to-severe COPD. N Engl J Med. 2014 Jun 5;370(23):2201-10. doi: 10.1056/NEJMoa1403086. Epub 2014 May 18. PMID 24836125

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 433 | 452
Completed | 386 | 397
Not Completed | 47 | 55
Not completed — Withdrawal by Subject | 16 | 20
Not completed — Lost to Follow-up | 3 | 5
Not completed — Death | 28 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Placebo | Total
Number analyzed (Participants) | 433 | 452 | 885
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.5) | 62.3 (8.4) | 62.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 203 | 387
  Male | 249 | 249 | 498
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 429 | 445 | 874
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 99 | 91 | 190
  White | 328 | 346 | 674
  More than one race | 2 | 11 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 362 | 376 | 738
  Canada | 71 | 76 | 147
Smoking History (Pack Years) [Mean (Standard Deviation); unit: Pack Years] | 50.0 (26.1) | 51.2 (28.7) | 50.6 (27.4)
Post-bronchodilator FEV1 (forced expiratory volume at one second) [Mean (Standard Deviation); unit: liters (L)] | 1.19 (0.58) | 1.19 (0.56) | 1.19 (0.57)
FEV1/FVC (forced expiratory volume at one second/forced vital capacity) [Mean (Standard Deviation); unit: Ratio] | 0.44 (0.13) | 0.44 (0.13) | 0.44 (0.13)
FEV1 (% Predicted) [Mean (Standard Deviation); unit: percent predicted] | 41.5 (17.8) | 41.6 (17.6) | 41.6 (17.7)
Acute COPD Exacerbation requiring Hospitalization or ED visit within previous 12 mo [Number; unit: participants] — Acute COPD (Chronic Obstructive Pulmonary Disease) Exacerbation requiring Hospitalization or Emergency Department visit within previous 12 months
  participants
    Yes | 216 | 238 | 454
    No | 217 | 214 | 431
Systemic glucocorticoid or antibiotic use within previous 12 mo [Number; unit: participants]
  Yes | 367 | 382 | 749
  No | 66 | 70 | 136
Use of supplemental oxygen within previous 12 mo [Number; unit: participants]
  Yes | 198 | 222 | 420
  No | 235 | 230 | 465

OUTCOME MEASURES:

1. Primary Outcome: Rates of COPD Exacerbations
Time Frame: up to 37 months
Population: Analysis excludes participants without any follow-up data.
Measure: Mean (Standard Deviation); unit: exacerbations/person-year
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 430 | 447
exacerbations/person-year | 1.36 (1.61) | 1.39 (1.73)
Statistical Analysis 1: Comparison: Simvastatin vs Placebo; Test type: Superiority or Other; p = 0.54, negative binomial regression; Adjustments of confidence intervals for between-participant variation (overdispersion)

2. Secondary Outcome: Time to First COPD Exacerbation
Time Frame: up to 37 months
Population: Analysis excludes participants without any follow-up data.
Measure: Median (95% Confidence Interval); unit: Days to the first exacerbation
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 430 | 447
Days to the first exacerbation | 223 [195 to 275] | 231 [193 to 303]
Statistical Analysis 1: Comparison: Simvastatin; Test type: Superiority or Other; p = 0.34, Log Rank

3. Secondary Outcome: Change in FEV1 (% Pred) From Baseline to Last Measure
Time Frame: Baseline, last measure at up to 37 months
Population: Analysis excludes participants without any follow-up data.
Measure: Median (90% Confidence Interval); unit: percent predicted
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 356 | 356
percent predicted | -0.86 [-11.04 to 8.67] | -1.81 [-10.62 to 7.10]
Statistical Analysis 1: Comparison: Simvastatin vs Placebo; Test type: Superiority or Other; p = .1461, t-test, 2 sided

4. Secondary Outcome: Acute Exacerbation COPD Hospitalization Rates (Events/Patient Year)
Time Frame: up to 37 months
Population: Analysis excludes participants without any follow-up data.
Measure: Mean (95% Confidence Interval); unit: events per patient year
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 430 | 447
events per patient year | 0.31 [0.24 to 0.38] | 0.31 [0.23 to 0.38]

ADVERSE EVENTS:
Time Frame: Up to 37 months
Arm/Group | Simvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 178/433 | 190/452
Other Adverse Events (participants affected / at risk) | 316/433 | 329/452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=433) | Placebo (N=452)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Other Infection (Infections and infestations) | 0 (0) | 1 (1) — Pulmonary Aspergillosis
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Respiratory Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (12) | 10 (14)
Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Genitourinary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 5 (7)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metabolic disorders (Metabolism and nutrition disorders) | 5 (6) | 5 (5)
Cavernous Hemangioma (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Mental Disorder (Psychiatric disorders) | 3 (4) | 5 (6)
Central Nervous System disorders (Nervous system disorders) | 1 (1) | 0 (0)
Pain (Nervous system disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Orbital cellulitis (Eye disorders) | 0 (0) | 1 (1)
Rheumatic Heart Disease (Cardiac disorders) | 1 (1) | 0 (0)
Ischemic Heart Disease (Cardiac disorders) | 4 (4) | 6 (6)
Pulmonary Circulation disorders (Cardiac disorders) | 4 (5) | 6 (6)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Dysrhythmias (Cardiac disorders) | 7 (7) | 4 (5)
Heart Failure (Cardiac disorders) | 4 (6) | 5 (7)
Cerebrovascular (Vascular disorders) | 1 (1) | 6 (6)
Artery disorder (Vascular disorders) | 2 (2) | 2 (3)
Vein disorder (Vascular disorders) | 4 (4) | 3 (4)
Acute Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 34 (40) | 27 (32)
Influenza (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (9)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumoconioses (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 96 (155) | 97 (187)
COPD other (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 10 (15)
Other Respiratory (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 13 (20)
Esophagus and stomach disorders (Gastrointestinal disorders) | 1 (1) | 5 (5)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Enteritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Other Intestinal disorders (Gastrointestinal disorders) | 7 (9) | 5 (5)
Other Digestive Disorders (Gastrointestinal disorders) | 11 (14) | 7 (8)
Nephrotic disorders (Renal and urinary disorders) | 2 (2) | 0 (0)
Other Urinary Disorder (Renal and urinary disorders) | 5 (5) | 5 (5)
Disorders of the Male Genitourinary System (Renal and urinary disorders) | 0 (0) | 2 (3)
Disorders of the Female Genitourinary System (Renal and urinary disorders) | 1 (1) | 1 (1)
Skin Infection (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Dorsopathy (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Rheumatism (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteopathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Nissen Fundoplication (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (General disorders) | 5 (5) | 1 (1)
Dizziness (General disorders) | 2 (2) | 0 (0)
Severe Headaches (General disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ill defined abdominal pain (General disorders) | 2 (2) | 3 (4)
Sudden death of unknown cause (General disorders) | 4 (4) | 4 (4)
Fractures (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Intracranial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Internal Injury (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Trauma from motorcycle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Complications of surgical and medical care (General disorders) | 4 (4) | 2 (2)
Respiratory Arrest (General disorders) | 2 (2) | 1 (1)
Abnormal Gait (General disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Degenerative Disc Disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Sepsis (General disorders) | 1 (1) | 4 (4)
Ill Defined Respiratory events (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 13 (15)
Ill defined digestive symptoms (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=433) | Placebo (N=452)
Acute Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 109 (159) | 107 (166)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 17 (19)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 232 (642) | 244 (649)
Other COPD Related Symptoms (Respiratory, thoracic and mediastinal disorders) | 41 (79) | 43 (80)
Arthropathies (Musculoskeletal and connective tissue disorders) | 25 (38) | 32 (43)
Dorsopathies (Musculoskeletal and connective tissue disorders) | 27 (35) | 27 (32)
Rheumatism (Musculoskeletal and connective tissue disorders) | 67 (89) | 54 (73)
Urinary Infection (Renal and urinary disorders) | 26 (56) | 23 (30)
Headache (General disorders) | 16 (20) | 23 (27)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 65 (94) | 59 (90)

LIMITATIONS AND CAVEATS:
Early termination by the Data and Safety Monitoring Board due to futility in respect to a treatment effect. The original study population goal was 1200 and the study was terminated at 885 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No